CLINICAL TRIAL: NCT04727736
Title: Phase 2 Study of 18F-DCFPyL Positron Emission Tomography (PET) in Men With Intermediate or High Risk Biochemically Recurrent Prostate Cancer
Brief Title: 18F-DCFPyL Positron Emission Tomography (PET) in Intermediate or High Risk Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Intervention became FDA-approved
Sponsor: Ashok Muthukrishnan (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ashok Muthukrishnan, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCC 20-009
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL + PET imaging (Experimental): Participants will receive a single dose of 18F-DCFPyL and undergo a PET imaging study.
  (The PET imaging may be repeated at a later date if the biopsy of the lesion is negative and if the lesion is present on follow-up imaging.)
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — 18F-DCFPyL (single dose injection) - a radiolabeled prostate-specific membrane antigen (PSMA) ligand

SUMMARY:
This is an interventional, single group assignment, prospective nonrandomized, open label Phase 2 trial designed to evaluate 18F-DCFPyL PET imaging in men diagnosed with prostate cancer with increasing prostate-specific antigen (PSA) levels.

DETAILED DESCRIPTION:
This is an trial designed to evaluate the positive predictive value of 18F-DCFPyL PET imaging in men diagnosed with prostate cancer with increasing PSA levels. Patients will receive a single dose of 18FDCFPyL PET and undergo a PET imaging study. 18F-DCFPyL Injection is an 18F-labeled small molecule that targets the extracellular domain of PSMA. One intravenous catheter will be placed for radiopharmaceutical administration. Patients will be injected with ≤ 333 MBq (≤ 9 mCi) of 18F-DCFPyL via this catheter. The dose range for 18F-DCFPyL will be 7 - 9 mCi. The PET imaging may be repeated at a later date if the biopsy of the lesion is negative and if the lesion is present on follow-up imaging.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer
* Biochemical recurrence was defined as a PSA of 0.2 or more ng/mL measured more than 6 weeks after prostatectomy or a PSA of 2 or more ng/mL rise above nadir following radiation therapy (ASTRO Phoenix consensus definition)
* Age ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Ability to understand and willingness to sign a written informed consent document
* Willing to comply with clinical trial instructions and requirements

Exclusion Criteria:

* History of another active malignancy within 3 years, other than basal cell and squamous cell carcinoma of the skin
* Presence of prostate brachytherapy implants unless approved by the PI
* Administration of another radioisotope within five physical half-lives of trial enrollment
* Radiation or chemotherapy within 2 weeks prior to trial enrollment
* Estimated glomerular filtration rate (eGFR) < 15 ml/mmol
* Serum total bilirubin > 3 times the upper limit of normal
* Aspartate transaminase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal
* Inadequate venous access
* Claustrophobia or any other condition that would preclude PET imaging
* Patients must not be receiving ADT except per criteria directly below. Patients who received in the past must have a serum testosterone that is recovered to at least 100 ng/dL.
* Patients who have been on ADT +/- novel hormonal agent (NHA) and developed M0 CRPC

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Intermediate or High Risk Biochemically Recurrent Prostate Cancer
Enrollment: 47 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Muthukrishnan, MD, MS, Principal Investigator — University of Pittsburgh - Associate Professor
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-DCFPyL + PET Imaging: Participants will receive a single dose of 18F-DCFPyL and undergo a PET imaging study.
  (The PET imaging may be repeated at a later date if the biopsy of the lesion is negative and if the lesion is present on follow-up imaging.)
  18F-DCFPyL: 18F-DCFPyL (single dose injection) - a radiolabeled prostate-specific membrane antigen (PSMA) ligand
Period: Overall Study
Arm/Group | 18F-DCFPyL + PET Imaging
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients that received study intervention and were radiologically evaluable.
Arm/Group | 18F-DCFPyL + PET Imaging
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 67 [65 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Positive Predictive Value (PPV) (Per-patient)
Description: Number of patients with true positive scans (TP - positive test with disease) divided by number of TP plus number of false positive scans (FP - positive test without disease). A scan will be deemed 'positive' if at least one lesion suggestive of disease recurrence is noted. Prostate lesions and lymph nodes will be considered positive if the uptake in those lesions exceeds blood pool activity. Bone lesions will be recorded as positive if the activity is higher than normal bone marrow uptake.
Time Frame: Up to 12 months
Population: Male patients diagnosed with prostate cancer with increasing PSA levels.
Measure: Number (95% Confidence Interval); unit: Per-patient percentage
Arm/Group | 18F-DCFPyL + PET Imaging
Number analyzed (Participants) | 47
Per-patient percentage | 83.9 [66.3 to 94.5]

2. Secondary Outcome: Positive Predictive Value (PPV) (Per-region)
Description: Number of true positive scans (TP - positive test with disease) divided by number of TP plus number of false positive scans (FP - positive test without true disease), by region (prostate bed, locoregional lymph nodes, distant lymph nodes, bones, and/or visceral organs). A scan will be deemed 'positive' if at least one lesion suggestive of disease recurrence is noted. Prostate lesions and lymph nodes will be considered positive if the uptake in those lesions exceeds blood pool activity. Bone lesions will be recorded as positive if the activity is higher than normal bone marrow uptake.
Time Frame: Up to 12 months
Population: Male patients diagnosed with prostate cancer with increasing PSA levels.
Measure: Number (95% Confidence Interval); unit: percentage per anatomical region
Arm/Group | 18F-DCFPyL + PET Imaging
Number analyzed (Participants) | 47
percentage per anatomical region
  In prostate bed | 50 [6.8 to 93.2]
  In LN pelvis | 96 [79.6 to 99.9]
  In LN extra-pelvis | 80 [28.4 to 99.5]
  In bone lesions | 85.7 [42.1 to 99.6]

ADVERSE EVENTS:
Time Frame: Patient observed for 1 year after they received the intervention.
Description: No AEs or SAEs were reported per CTCAE v4.0.
Arm/Group | 18F-DCFPyL + PET Imaging
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT04727736/Prot_SAP_000.pdf